CLINICAL TRIAL: NCT02423408
Title: A Proof-of-Concept Phase 2, Double-Blind, Randomized, Multicenter, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TNX-201 for the Treatment of A Single Tension-Type Headache
Brief Title: Safety and Efficacy Study of TNX-201 Capsules for Treatment of Single Tension-Type Headache
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-IS-T201
Record Dates: First submitted 2015-04-15; First posted 2015-04-22 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2016-12

CONDITIONS: Tension-Type Headache
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TNX-201 (Experimental): 4 X 35 mg capsules to be taken when qualifying tension-type headache occurs
  Interventions: Drug: TNX-201
- Placebo (Placebo Comparator): 4 X placebo capsules to be taken when qualifying tension-type headache occurs
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TNX-201 — TNX-201 capsule
  Other Names: (R)-isometheptene mucate
  Arms: TNX-201
Drug: Placebo — Placebo capsule
  Other Names: TNX-201 Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, multicenter, double-blind, placebo-controlled, parallel-group study to evaluate the safety and efficacy of a single dose of TNX-201 (140 mg) for the treatment of a single qualifying Tension-Type-Headache (TTH).

DETAILED DESCRIPTION:
The study will be conducted in 4 periods (the Screening Period, the Run-In Period, the Double-Blind Treatment Period and the Follow-up Period) and 4 visits (the Screening Visit, Enrollment Visit, Randomization Visit and End-of-Study Visit).

Screening Period- Eligible subjects who provide written informed consent to participate will have study assessments performed at the Screening.

Run-In Period- The Run-In Period will last for at least 28 days. During the Run-In period, subjects will be assessed for frequency of headache, study compliance and to ensure they meet all required study criteria for randomization.

Double-Blind Treatment Period- The Double-Blind Treatment Period (Treatment Period) will last up to 4 weeks or until a qualifying headache episode has occurred and been treated using the study drug, whichever occurs first.

Follow-up Period- All subjects will return to the investigational site for this visit, regardless of whether they have treated a qualifying TTH with study medication. Subjects who have not treated a qualifying TTH with study drug during the Treatment Period will be asked to return study materials and undergo safety evaluations at the End-of-Study Visit and will be discharged from the study. Subjects who have treated a qualifying TTH with study drug during the Treatment Period will ingest a 140 mg dose of open-label TNX-201 at this visit and undergo urine and blood sample collection for 3 hours post-dose to characterize each subject's genetic metabolism and PK profile.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of reading and understanding English and able to provide written informed consent to participate.
2. Male or female adults ≥ 18 and < 65 years of age at the time of Visit 1.
3. Body mass index (BMI) ≥ 18.5 and ≤ 45.0.
4. Greater than 1 year history of episodic tension-type headache with onset prior to 50 years of age.
5. History of tension-type headaches that typically last ≥ 4 hours if untreated.
6. History of 2-14 tension-type headaches per month for the last 3 months prior to Visit 1.
7. Diagnosis must comply with the International Headache Society (IHS) diagnostic criteria.
8. No significant ECG findings at Screening
9. If female, is either not of childbearing potential or is practicing a predefined medically acceptable method of birth control (hormonal methods, intrauterine device, double-barrier method, sexually-exclusive vasectomized male partner, same-sex relationship) throughout the study.
10. Willing and able to comply with all protocol-specified requirements.

Exclusion Criteria:

1. Known or suspected hypersensitivity to isometheptene mucate or any excipients used in the formulation.
2. Use of any excluded concomitant medications.
3. Current use of opiate analgesics.
4. Use of any prophylactic drug therapy for headache control within 4 weeks of screening (e.g., anticonvulsants, mood stabilizers, beta-blocker, antidepressants, muscle relaxants, botulinum toxin). Subjects taking any of these medications for an indication other than headache (e.g., a beta-blocker for hypertension) will require medical monitor's approval prior to initiation of the Run-In Period.
5. History of medication use for acute headache on ≥ 10 days per month on average during the 3 months prior to Visit 1.
6. Positive results for addictive substances (e.g., cocaine, phencyclidine (PCP), amphetamines, opiates) at Screening.
7. History of migraine that exceeds a mean of four attacks per month during the preceding calendar year.
8. Lifetime history of schizophrenia, schizoaffective disorder, bipolar I/II disorder, delusional disorder, or psychotic disorder not otherwise specified.
9. Chronic pain disorders requiring medical treatment with opioids, chronic daily use of NSAIDs at the time of screening
10. History of coronary artery disease, coronary vasospasm, aortic aneurysm, peripheral vascular disease or other ischemic diseases (e.g., ischemic bowel syndrome or Raynaud's syndrome).
11. Inadequately controlled hypertension or persistently elevated systolic blood pressure or diastolic blood pressure upon repeat assessment at screening or on the day of randomization.
12. Current history of two or more CAD risk factors at Screening (tobacco use, receiving anti-hypertensive medication for hypertension, high LDL cholesterol or low HDL cholesterol levels, family history of premature CAD, diabetes mellitus)
13. History cerebral vascular accident, transient ischemic attack, seizure disorders.
14. Other clinically significant cardiac disease.
15. History of concurrent illness that requires hospitalization within 30 days prior to Visit 1.
16. Current evidence of human immunodeficiency virus infection or clinically significant hepatitis B or C infection.
17. Clinically significant laboratory abnormalities based on screening laboratory tests and/or medical history.
18. Participation in another investigational trial during the 30 days prior to Visit 1 or during this trial. Subjects who have participated in non-interventional trials may be permitted to participate on a case-by-case basis after review with the Medical Monitor.
19. Women who are pregnant, breast-feeding, or planning to become pregnant during this trial.
20. Any other household member currently participating in a Tonix-sponsored study or family member or relative of investigative staff.
21. Any condition and/or medical history that would make the subject unsuitable for study participation and completion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracie Ruther, M.S, Study Director — 1 513 579 9911 ext 2214
Locations (10):
- United States (10):
  - James D. Wolfe, MD, San Jose, California
  - Avail Clinical Research LLC., DeLand, Florida
  - Nathan Segall, MD, CPI, Stockbridge, Georgia
  - Michigan Head-Pain Neurological Institute, Ann Arbor, Michigan
  - Gary D. Berman, MD, Minneapolis, Minnesota
  - John Rubino, MD, Raleigh, North Carolina
  - PMG Research of Winston-Salem, LLC., Winston-Salem, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Stephan C. Sharp, MD, Nashville, Tennessee
  - Duane G. Wombolt, MD, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- TNX-201: 4 X 35 mg capsules to be taken orally with a minimum of 4 ounces of water when qualifying tension-type headache occurs
  TNX-201: TNX-201 capsule
- Placebo: 4 X placebo capsules to be taken orally with a minimum of 4 ounces of water when qualifying tension-type headache occurs
  Placebo: Placebo capsule
Period: Overall Study
Arm/Group | TNX-201 | Placebo
Started | 83 | 82
Completed | 82 | 80
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TNX-201 | Placebo | Total
Number analyzed (Participants) | 83 | 82 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 83 | 82 | 165
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 74 | 148
  Male | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Pain Free
Description: Number of subjects pain free at 2 hours post-dose (Pain assessed by 4-point NRS, VAS, and binary yes/no question).
  4-point NRS grades: 0=none, 1=mild, 2=moderate, 3=severe; "pain-free" defined as score = 0.
  VAS: 0-100 scale, anchored by verbal anchors of No Pain (0) vs. Worst Imaginable Headache Pain (100). "Pain-free" was defined as a score <= 5
Time Frame: 2 hours
Population: LOCF Analysis
  8 subjects in the TNX-201 group and 10 subjects in the placebo group who did not take a dose during the double-blind treatment period and/or did not report data 2-hour post-dose were excluded from analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | TNX-201 | Placebo
Number analyzed (Participants) | 75 | 72
Participants
  Binary Response | 21 | 20
  4-Point NRS | 21 | 19
  VAS | 20 | 21

2. Secondary Outcome: Number of Subjects Pain Free at 15, 30, 60, 90 Minutes and 4 Hours Post-dose (Pain Will be Assessed by 4-point NRS, VAS, and Binary Yes/no Question)
Description: 4-point NRS grades: 0=none, 1=mild, 2=moderate, 3=severe.
  VAS: 0-100 scale, No Pain vs. Worst Imaginable Headache Pain
Time Frame: 15, 30, 60, 90 minutes and 4 hours post-dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TNX-201 | Placebo
Number analyzed (Participants) | 75 | 72
Participants
  Binary Response : 15 Minutes | 1 | 0
  Binary Response : 30 Minutes | 4 | 2
  Binary Response : 60 Minutes | 9 | 8
  Binary Response : 90 Minutes | 13 | 17
  Binary Response : 4 Hours | 37 | 37
  4-Point NRS : 15 Minutes | 1 | 0
  4-Point NRS : 30 Minutes | 3 | 1
  4-Point NRS : 60 Minutes | 8 | 7
  4-Point NRS : 90 Minutes | 13 | 14
  4-Point NRS : 4 Hours | 37 | 35
  VAS : 15 Minutes | 2 | 0
  VAS : 30 Minutes | 4 | 2
  VAS : 60 Minutes | 8 | 5
  VAS : 90 Minutes | 13 | 13
  VAS : 4 Hours | 39 | 34

3. Secondary Outcome: Number of Subjects Using Rescue Medication During the 24-hour Post-dose Period
Time Frame: 24-hour post-dose period
Population: 8 subjects in the TNX-201 group and 10 subjects in the placebo group who did not take a dose during the double-blind treatment period and/or did not report data 2-hour post-dose were excluded from analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | TNX-201 | Placebo
Number analyzed (Participants) | 75 | 72
Participants | 16 | 15

4. Secondary Outcome: Number of Subjects With at Least a Two-category Improvement From Baseline at 2 Hours Post-dose in VAS Severity Category (Carvalho Responders)
Description: The Carvalho Responder analysis refers to subjects with at least 2 categories of improvement in their VAS severity category (0-100 scale). VAS severity categories were defined as "severe" if between 52-100 inclusive, "moderate" between 31-51 inclusive, "mild" between 6-30 inclusive, and pain-free if less than 6. Therefore, a Carvalho responder was either a subject who had a VAS response classified as 'severe' at baseline and 'mild' or pain-free at the post-dose assessment time point, or a subject who had a VAS response classified as 'moderate' at baseline and pain-free at the post-dose assessment time point.
Time Frame: 2 hours
Population: Only subjects who were categorized as "severe" or "moderate" at baseline and have data reported at 2 hours were included in this analysis. All subjects who took rescue medication at or before 2 hours were considered non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | TNX-201 | Placebo
Number analyzed (Participants) | 56 | 60
Participants | 24 | 24

ADVERSE EVENTS:
Description: 5 subjects in the TNX-201 group and 9 subjects in the placebo group did not take a dose of study drug during the double-blind treatment period; therefore, these subjects were not included in the analyses.
Arm/Group | TNX-201 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/73
Other Adverse Events (participants affected / at risk) | 5/78 | 6/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TNX-201 (N=78) | Placebo (N=73)
Dizziness (Nervous system disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Feeling Hot (General disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA in place with all study investigators.